CLINICAL TRIAL: NCT02229201
Title: Phase 1 Study of the Impact of Propofol vs. Sevoflurane on Brain Damage and Inflammatory Response During Brain Tumour Surgery
Brief Title: Comparison of Two Anaesthetics on Brain During Brain Tumour Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jasmina Markovic Bozic, MD, MSC, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCL-NKG-01
Record Dates: First submitted 2014-08-11; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Inflammation
Keywords: propofol; sevoflurane; Interleukin 6; Interleukin 10
MeSH Terms: conditions — Inflammation | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Experimental): intravenous anaesthetic
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): volatile anaesthetic
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — 4-6 mg/kg/h during anaesthesia
  Other Names: Propoven 1%
  Arms: Propofol
Drug: Sevoflurane — 0.8 MAC
  Other Names: Sevorane
  Arms: Sevoflurane

SUMMARY:
Anaesthesia and surgical stress during craniotomy can lead to brain damage and activation of inflammatory response. Consequently inflammatory cytokines (IL6, IL8, IL10) are released. Cell mediated immune balance can increase postoperative complications (infections, wound healing, multiple organ dysfunction). Many studies have shown that volatile anaesthetics reduce systemic and local inflammatory response during major surgery, but animal studies have shown that volatile anaesthetics can induce neuroinflammation (IL6, NF-κB) that leads to decline of cognitive function in rodent and possible human.

Our aim was to investigate how anaesthetic technique for craniotomy influences the release of inflammatory cytokines. Our hypothesis was that when optimal neuroprotective strategies are followed during surgery intravenous anaesthesia attenuates inflammatory response comparing to inhalational anaesthesia.

The investigators included 40 patients anaesthetised with remifentanil based anaesthesia with sevoflurane (S group) or propofol (P group).

Plasma levels of IL6, IL8, IL10 were measured during preoperative, perioperative and postoperative periods of both groups of patients. The investigators also noted emergence parameters, postoperative (pain, shivering, vomiting) and neurological complications after surgery.

DETAILED DESCRIPTION:
Anaesthetic technique for craniotomy has to provide optimal cerebral perfusion, oxygenation and prevent brain oedema (1). It also has to lower the stress response on pain during intubation and surgical manipulation. Emergence from anaesthesia has to be rapid and smooth to permit early postoperative neurological evaluation. The most likely opioid in the last decade is short acting opioid remifentanil that can be easy titrated during the procedure and provides early recovery (2, 3, 4, 5). Currently the propofol-remifentanil and sevoflurane-remifentanil are the most frequently used combinations for craniotomy (6, 7). Recently a multicentre study was published that did not show differences in early recovery between three groups (propofol-remifentanil: TIVA, sevoflurane-remifentanil, sevoflurane-fentanyl). Either technique provided optimal surgical conditions. The group received TIVA had attenuated changes in stress biomarkers (cortizol in plasma and urine, cateholamines. (8).

Anaesthesia and surgical stress during craniotomy can lead to brain damage and activation of inflammatory response (9, 10). Consequently inflammatory cytokines (IL6, IL8, IL10) are released. Cell mediated immune balance can increase postoperative complications (infections, wound healing, multiple organ dysfunction). Many studies have shown that volatile anaesthetics reduce systemic and local inflammatory response during major surgery (11, 12, 13, 14), but animal studies have shown that volatile anaesthetics can induce neuroinflammation (IL6, NF-κB) that leads to decline of cognitive function in rodent and possible human (15,16).

Our aim was to investigate how anaesthetic technique for craniotomy influences the release of inflammatory cytokines. Our hypothesis was that when optimal neuroprotective strategies are followed during surgery intravenous anaesthesia attenuates inflammatory response comparing to inhalational anaesthesia.

Plasma levels of IL6, IL8, IL10 were measured during preoperative, perioperative and postoperative periods of both groups of patients. The investigators also noted emergence parameters, postoperative (pain, shivering, vomiting) and neurological complications after surgery.

Patients and methods

Anaesthesia regimen:

On arrival in the operating room, the patients were randomly assigned to either Group P or Group S. Randomisation was done according to computer-generated order.

All patients were on a regimen of dexamethasone 4x4mg/day with the first dose given at least one day before surgery.

After arriving to the operating room the standard monitoring was instituted. An arterial catheter was placed in the radial artery to continuously monitor blood pressure. For extended haemodynamic monitoring Vigileo system was used.

Patients were premedicated with midazolam (2-3 mg i.v.) and ondansetron (4-8 mg i.v.). Antibiotic prophylaxis with intravenous cefazolin 2g/100 ml 0.9% NaCl was invariably used in all patients.

Anaesthesia induction in Group P was performed with propofol (Propoven, Fresenius Kabi) and in Group S with sevoflurane (Sevorane, Abbott Laboratories). Before intubation all patients received remifentanil (Ultiva, GlaxoSmithKline) and rocuronium (Esmeron, MSD).

After intubation, patient's lungs were ventilated mechanically, with 1:2 oxygen-air mixtures in P and S group. Ventilation was adjusted to maintain normocapnia. Anaesthesia was maintained by continuous infusion of propofol 4-6 mg/kg/h in the P group and with sevoflurane 0,8-1 MAC in the S group. Remifentanil was adjusted regarding to anaesthesia response (0.1 - 2 μg/kg/min). The depth of anaesthesia was measured by a bispectral index (BIS) monitor; BIS values were maintained at 40-60.

For haemodynamic management the following algorithm was used: continuous infusion of 0.9% NaCl 6 mL kg-¹ for the first hour, followed by 2.5 ml kg-¹h-¹ . If CI < 2 L/min/m2and SVV > 10%, 6% hydroxyethyl starch (Voluven, Fresenius Kabi) until SVV-10% ; if there is no improvement after 250 ml 6% HES-a, ephedrine (0.5% Efedrin, UMC Ljubljana Pharmacy) 5-10 mg iv or fenilefrin 50-100 μg (0.01%, UMC Ljubljana Pharmacy). If CI < 2 L/min/m2, SVV < 10% and heart beat < 40/min, atropine 0,5 mg. If the mean arterial pressure increases by more than 30% and the heart rate by more than 30% from baseline, the infusion of remifentanil is increased. Any adverse hemodynamic events that did not respond to changes in anaesthetic regimen could be managed with urapidil or metoprolol, as appropriate. Hypotension following blood losses was maintained with colloids (6% HAES) and blood replacement. Hemodynamic parameters were monitored continuously at 5-min intervals from the beginning of induction until the patients were discharged from the PACU.

30 minutes before the end of the surgery (at the time of dura closer) piritramid 5-10 mg was administered. Continuous intravenous infusion of piritramid was started postoperatively as patient control analgesia (PCA). The time of the operation was determined as the time from pin head-holder placement to its removal. The time from the end of the operation to the tracheal extubation was also noted. All patients were extubated in the operating theatre and then transferred to the recovery room.

Postoperative management:

After surgery, the patients stayed in the recovery room for one hour and were then transferred to the intensive care unit of the Department of Neurosurgery.

Standard postoperative monitoring generally used in these procedures was implemented. Oxygen titrated to the lowest level needed to achieve the target arterial oxygen saturation of 96%, was administered via a Venturi mask. Post anaesthetic adverse events and medication in ICU were recorded for a period of 24 h after anaesthesia. Adverse events were defined as any unintended changes in body function or well being, such as hypertension, postoperative nausea and vomiting, pain, neurological complications, in particular if clinical intervention or drug therapy was required.

Hospital stay was also recorded.

Study design:

This prospective randomised single centre study was conducted at the Department of Anaesthesiology and Surgical Intensive Care and at the Department of Neurosurgery, in close cooperation with the Department of Clinical Chemistry and Biochemistry, University Medical Centre Ljubljana. The investigators included 40 patients anaesthetised with remifentanil based anaesthesia with sevoflurane (S group) or propofol (P group). The study was approved by the National Medical Ethics Committee of the Republic of Slovenia. All the procedures were performed in accordance with Helsinki declaration. The written informed concern was obtained from all included patients. The patients included in the study were given anaesthesia by the same anaesthesiologist.

The data recorded included demographic characteristics, time of surgery, time to extubation, hemodynamic parameters.

Arterial blood samples for the determinations of cytokines (IL 6, IL 8, IL 10) were drawn at the following time points: 1. before induction, 2. During tumor resection 3. at the end of the surgery, and 4. 24 hours after surgery 5. 48 hours after surgery.

For analyses of serum interleukin-6 (IL-6), interleukin-8 (IL-8) and interleukin-10 (IL-10), blood samples were collected in tubes without additive. After centrifugation serum samples were stored at -20 ºC until analysis. Analyses of samples were performed in one batch. Chemiluminescent immunometric assay (Immulite analyzer; Siemens Healthcare, Erlangen, Germany) was used to measure the concentrations of IL-6, IL-8, and IL-10.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* American Society of Anaesthesiologists (ASA) physical status I-III
* Scheduled for brain tumour surgery
* Glasgow Coma Score 15
* Cooperative

Exclusion Criteria:

* No written informed consent
* Eendocrine systematic disease
* Ddrugs that alter endocrine metabolism
* History of drug hypersensitivity
* Drug addiction
* Perioperative blood derivatives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Interleukin 10 plasma concentrations | Within 48 hours (1. Before surgery and anaesthesia 2. During surgery, 3. At the end of surgery 4.First postoperative day 5.Second postoperative day)
  The interleukin 10 plasma concentrations during craniotomy (preoperative, perioperative and postoperative periods)

SECONDARY OUTCOMES:
Hospital stay | within the first 15 days after surgery
Pulmonary complications | within the first 15 days after surgery
Cardiovascular complications | within the first 15 days after surgery
Neurological complications | within the first 15 days after surgery
Reoperation | within the first 15 days after surgery
Death | within the first 15 days after surgery
Postoperative nausea and vomiting (PONV) | within the first 24 hours after surgery
  Post anaesthetic adverse events and medication in ICU were recorded for a period of 24 h after anaesthesia. Adverse events were defined as any unintended changes in body function or well being.
Pain using VAS score | within the first 24 hours after surgery
  Post anaesthetic adverse events and medication in ICU were recorded for a period of 24 h after anaesthesia. Adverse events were defined as any unintended changes in body function or well being, in particular if clinical intervention or drug therapy was required.
Change of blood pressure from the baseline | within the first 24 hours after surgery
  Post anaesthetic adverse events and medication in ICU were recorded for a period of 24 h after anaesthesia. Adverse events were defined as any unintended changes in body function or well being, in particular if clinical intervention or drug therapy was required.

OTHER OUTCOMES:
Consumption of Propofol (mg) | within first 12 hours from the time before the surgery until the end of surgery
  Drugs consumption, volume loading, blood loss and post anaesthetic adverse events and medication were recorded:
Consumption Remifentanil (mg) | within first 12 hours from the time before the surgery until the end of surgery
  Drugs consumption, volume loading, blood loss and post anaesthetic adverse events and medication were recorded.
Consumption of efedrin (mg) | within first 12 hours from the time before the surgery until the end of surgery
  Efedrin was used for correction of low blood pressure
Total loss of blood (ml) | within first 12 hours from the time before the surgery until the end of surgery
Time to extubation (min) | within first 12 hours from the end of surgery until release from the recovery room
  Post anaesthetic adverse events and medication:
Vomiting (yes/no) | within first 12 hours from the end of surgery until release from the recovery room
  Post anaesthetic adverse events and medication:
Lowering of arterial pressure (yes/no) | within first 12 hours from the end of surgery until release from the recovery room
  Post anaesthetic adverse events and medication:
Additional piritramid (yes/no) | within first 12 hours from the end of surgery until release from the recovery room
  Post anaesthetic adverse events and medication:
Consumption of fenilefrin (mikrog) | within first 12 hours from the time before the surgery until the end of surgery
  Fenilefrin was used for low blood pressure correction
Volume loading (ml) | within first 12 hours from the time before the surgery until the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jasmina Markovic Bozic, MD, MSC, Principal Investigator — CD of Anaesthesiology and Intensive Therapy, University Medical Centre Ljubljan; Blaz Karpe, PHD, Principal Investigator — Faculty of Natural Science and Engineering, University of Ljubljana; Iztok Potocnik, MD, MSC, Principal Investigator — CD of Anaesthesiology and Intensive Therapy, University Medical Centre Ljubljan; Ales Jerin, PHD, Principal Investigator — CLINICAL INSTITUTE OF CLINICAL CHEMISTRY AND BIOCHEMISTRY, University Medical Centre Ljubljana; Andrej Vranič, MD, PHD, Principal Investigator — CD of Neurosurgery, University Medical Centre Ljubljana; Vesna Novak Jankovic, PROF, PHD, Study Chair — CD of Anaesthesiology and Intensive Therapy, University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Blum FE, Zuo Z. Volatile anesthetics-induced neuroinflammatory and anti-inflammatory responses. Med Gas Res. 2013 Aug 1;3(1):16. doi: 10.1186/2045-9912-3-16. PMID 23915963
- [Background] El Beheiry H. Protecting the brain during neurosurgical procedures: strategies that can work. Curr Opin Anaesthesiol. 2012 Oct;25(5):548-55. doi: 10.1097/ACO.0b013e3283579622. PMID 22895122
- [Derived] Markovic-Bozic J, Karpe B, Potocnik I, Jerin A, Vranic A, Novak-Jankovic V. Effect of propofol and sevoflurane on the inflammatory response of patients undergoing craniotomy. BMC Anesthesiol. 2016 Mar 22;16:18. doi: 10.1186/s12871-016-0182-5. PMID 27001425